CLINICAL TRIAL: NCT01281384
Title: Routine vs Selective Cardiac Magnetic Resonance in Non-Ischemic Heart Failure (OUTSMART-HF) Project I-B of Imaging Modalities to Assist With Guiding Therapy and the Evaluation of Patients With Heart Failure (IMAGE-HF)
Brief Title: Routine vs Selective Cardiac Magnetic Resonance in Non-Ischemic Heart Failure
Acronym: OUTSMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Principal Investigator, Rob Beanlands, Rob S. Beanlands, MD, FRCPC, Chief of Cardiology, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Project I-B; CIF-99470 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure
Keywords: cardiac magnetic resonance imaging; echocardiography; heart failure; imaging; cost effectiveness; quality of life; definitive diagnosis; prospective comparative effectiveness randomized clinical trial
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard imaging (echocardiography) (Active Comparator): Subjects will undergo their clinically indicated echocardiogram as ordered by their attending physician.
  Interventions: Other: Standard Imaging
- Advanced Imaging (Cardiac MRI) (Active Comparator): Subjects will undergo their clinically indicated echo as ordered by their attending physician, plus a cardiac MRI, which will be scheduled within 14 days of the echo.
  Interventions: Other: Advanced Imaging

INTERVENTIONS:
Other: Advanced Imaging
  Other Names: Cardiac Magnetic Resonance Imaging (CMR)
  Arms: Advanced Imaging (Cardiac MRI)
Other: Standard Imaging
  Other Names: Echocardiography
  Arms: Standard imaging (echocardiography)

SUMMARY:
Uncovering the underlying cause of heart failure can be quite challenging and doctors often rely on imaging tests such as echo (heart ultrasound) to provide the answers. Cardiac MRI is emerging as another promising test because it gives very precise information on heart function and the amount of scarring in the muscle. Heart failure patients are increasingly being sent for cardiac MRI but the potential advantage that this test offers over others such as echo has not been fully explored.

The purpose of this study is to determine if cardiac MRI provides more information on the cause of heart failure than traditional tests such as echo. In addition, if the information provided by this test always leads to an overall improvement in a patient's heart condition over time.

This is a randomized study where subjects referred for clinically indicated heart failure workup to determine the best clinical management will undergo standard heart failure testing (including echo) OR standard testing PLUS cardiac MRI.

DETAILED DESCRIPTION:
Primary objective: to compare the effect of routine cardiac magnetic resonance (CMR) versus standard care (i.e. echocardiography with only selective use of CMR) on the etiological diagnosis in patients with a non-ischemic heart failure (HF). The proposed categories of HF to be considered in this study include: idiopathic dilated cardiomyopathy, infiltrative cardiomyopathy, inflammatory, hypertrophic cardiomyopathy, heart failure with preserved ejection fraction (HFPEF), ischemic cardiomyopathy, mixed etiology and other (eg. pericardial, congenital, non-compaction, right ventricular failure).

Primary hypothesis: Routine use of CMR (vs. selective use) will lead to a more specific diagnostic characterization of the underlying etiology of non-ischemic heart failure. This will lead to a reduction in the diagnosis of idiopathic dilated cardiomyopathy and HFPEF.

Secondary objectives: Determine the effects that routine use of CMR in non-ischemic HF has on therapeutic decisions, on the Composite Clinical Endpoint (CCE), cardiac function, symptoms, quality of life (QoL), and costs. Ancillary measurements will include the safety of imaging tests and adverse reactions to gadolinium contrast agent.

Secondary hypothesis: Routine use of CMR will have significant impact on treatment decisions, (1) lead to more disease specific therapies and/or (2) cause a significant change in the number and class of HF meds, during follow-up. The routine CMR group will also have improved clinical outcomes (CCE), symptoms and QoL and decreased costs to the standard of care group during follow-up.

Design

Methods: Randomized controlled trial comparing i) routine CMR vs. ii) echocardiography with selective CMR in patient with HF due to NICM and/or HFPEF.

Among patients enrolled in Level I of IMAGE-HF, it is expected that 504 will have known NICM (or strongly suspected based on young age, absent risk factors and presenting history) and/or HFPEF.

Tertiary care sites (in Canada and Finland) with dedicated HF programs will participate in the study. Consecutive patients will be enrolled at sites with dedicated CMR programs (defined as minimum 200 cases/year and maximum 2 weeks waiting time in the majority of patients) and randomized to routine CMR or selective CMR. Non-ischemic HF patients from sites without dedicated CMR programs will be included in a registry of patients undergoing routine HF care (i.e. selective use of CMR). Participants in the selective CMR arm may ONLY undergo CMR for a suspicion of: 1) infiltrative myocardial disease, 2) arrhythmogenic right ventricular cardiomyopathy, 3) adult congenital heart disease or 4) pericardial disease following standard HF care including echocardiography. Other tertiary sites may be added in year 2-3 depending on recruitment needs and registry sites may become randomization sites if the experience and wait-time criteria are met.

ELIGIBILITY:
The study population includes patients with either

1. Newly diagnosed HF within the past 12 months

   OR
2. Established HF patients with deterioration/decompensation within the past 12 months

Inclusion Criteria: Patients with new or worsening HF as above AND

1. Age > 18
2. Working clinical diagnosis (known or highly suspected) of non-ischemic cardiomyopathy (NICM) OR Clinical diagnosis of HFPEF (Signs or symptoms of heart failure with a LVEF ≥ 40%)
3. Documented history of Class II-IV NYHA HF symptoms within the past 12 months

Exclusion Criteria:

1. Prior CMR and no major change in clinical condition
2. Well-documented specific etiology (eg known amyloidosis or hemochromatosis)
3. MD considers cause of heart failure is attributable to obstructive CAD.
4. Documented previous STEMI (any territory) or NSTEMI in LAD territory
5. Severe medical conditions that significantly affect the patient's outcome (eg. active malignancy)
6. Ongoing need for advanced cardiac life support (eg IABP)
7. Severe valvular heart disease requiring surgery within the next 6 months
8. Contraindications to CMR (e.g. certain metallic implants, severe claustrophobia)
9. Contraindications to gadolinium contrast agent (GFR < 30ml/min/1,72m2, pregnancy)
10. Inability to give informed consent
11. Evidence of multivessel ischemia on stress imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2011-01; Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of definitive diagnoses | 3 and 12 months
  Following the completion of all baseline testing (including echo) in the selective arm and baseline testing + CMR in the routine arm, the treating physician will assign a diagnosis on a standardized template using all available information. The diagnosis of non-ischemic cardiomyopathies will be based upon recent Canadian Consensus Statement.
  Expected Result - The routine CMR group will have a significantly higher rate of specific diagnoses for (a) heart failure with preserved systolic function (HFPSF) and (b) dilated cardiomyopathy (DCM) diagnoses (i.e. fewer idiopathic DCM) than the selective CMR group.

SECONDARY OUTCOMES:
Treatment effects | 3 and 12 months
  Telephone follow up will be conducted. The presence of each HF medication class will be re-assessed in addition to the overall number of cardiac medications. The presence of advanced HF therapies will additionally be recorded at each follow-up visit including: implantable device, electrophysiologic study/ablation, cardiac surgery/transplantation, and disease specific therapies (eg. phlebotomy for hemochromatosis; steroids for sarcoidosis). The HF specialist supervising the follow-up visits will also be asked to reassess the HF etiology during each encounter.
Clinical Endpoints | 3 and 12 months
  CCE (Death, Cardiovascular (CV) death, HF admission), left ventricular (LV) Function, QoL, Referral to HF clinic, Costs and Safety) will be assessed.
Resource utilization and costs | 3 and 12 months
  Regression methods will be used to assess the incremental costs associated with the routine use of CMR.
HF Diagnosis Variability: | 3 and 12 months
  A local independent blinded heart failure expert will also be asked to diagnose the HF etiology in a subset of 100 patients (~10%) in order to determine inter-observer variability in each of the CMR selective and standard arms.
Echo/CMR variability: | baseline
  An anonymized copy of each CMR and each available echo will be sent to a core lab. A second interpretation will occur at the core lab in 10% of cases in order to assess reproducibility and quality assurance of the results.

CONTACTS AND LOCATIONS:
Overall Officials: Rob SB Beanlands, MD, FRCP C, Study Director — Universityof Ottawa Heart Institute; Ian Paterson, MD, Principal Investigator — University of Alberta
Locations (14):
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - University of Laval, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
- Finland (3):
  - Helsinki University Central Hospital,, Helsinki
  - University of Kuopio, Kuopio
  - University of Turku, Turku

REFERENCES:
- [Background] Paterson DI, OMeara E, Chow BJ, Ukkonen H, Beanlands RS. Recent advances in cardiac imaging for patients with heart failure. Curr Opin Cardiol. 2011 Mar;26(2):132-43. doi: 10.1097/HCO.0b013e32834380e7. PMID 21297464
- [Background] Paterson I, Wells GA, Ezekowitz JA, White JA, Friedrich MG, Mielniczuk LM, O'Meara E, Chow B, DeKemp RA, Klein R, Dennie C, Dick A, Coyle D, Dwivedi G, Rajda M, Wright GA, Laine M, Hanninen H, Larose E, Connelly KA, Leong-Poi H, Howarth AG, Davies RA, Duchesne L, Yla-Herttuala S, Saraste A, Farand P, Garrard L, Tardif JC, Arnold M, Knuuti J, Beanlands R, Chan KL. Routine versus selective cardiac magnetic resonance in non-ischemic heart failure - OUTSMART-HF: study protocol for a randomized controlled trial (IMAGE-HF (heart failure) project 1-B). Trials. 2013 Oct 12;14:332. doi: 10.1186/1745-6215-14-332. PMID 24119686
- [Derived] Paterson DI, Wells G, Erthal F, Mielniczuk L, O'Meara E, White J, Connelly KA, Knuuti J, Radja M, Laine M, Chow BJW, Kandolin R, Chen L, Dick A, Dennie C, Garrard L, Ezekowitz J, Beanlands R, Chan KL; IMAGE-HF Investigators. OUTSMART HF: A Randomized Controlled Trial of Routine Versus Selective Cardiac Magnetic Resonance for Patients With Nonischemic Heart Failure (IMAGE-HF 1B). Circulation. 2020 Mar 10;141(10):818-827. doi: 10.1161/CIRCULATIONAHA.119.043964. Epub 2020 Jan 8. PMID 31910649